CLINICAL TRIAL: NCT05587257
Title: Transepidermal Drug Delivery of Minoxidil Via Either Fractional Carbon Dioxide Laser or Microneedling Versus Its Topical Nanoparticles Preparation for Treatment of Alopecia Areata
Brief Title: Role of Minoxidil in Alopecia Areata Transepidermal Drug Delivery of Minoxidil Via Either Fractional Carbon Dioxide Laser or Microneedling Versus Its Topical Nanoparticles Preparation for Treatment of Alopecia Areata
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Elsayed Mohamed, Assistant Lecturer, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Minoxidil in alopecia areata
Record Dates: First submitted 2022-10-16; First posted 2022-10-20 (Actual); Last update posted 2022-10-20 (Actual); Status verified 2022-10

CONDITIONS: Alopecia Areata
MeSH Terms: conditions — Alopecia Areata | interventions — Dosage Forms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1 (Experimental): six sessions of fractional carbon dioxide laser every 2 weeks will be done for 15 patients with alopecia areata followed immediately by topical application of minoxidil 5%
  Interventions: Device: Fractional CO2 laser
- Group 2 (Experimental): six sessions of microneedling evry 2 weeks will be done for 15 patients with alopecia areata followed immediately by topical application of minoxidil 5%
  Interventions: Device: Derma pen
- Group 3 (Experimental): 15 patient of alopecia areata that will be treated by topical nanominoxidil for 3 months.
  Interventions: Drug: Niosome minoxidil
- Group 4 (Active Comparator): 15 patient of alopecia areata that will be treated by topical minoxidil 5% for 3 months
  Interventions: Drug: Minoxidil Topical Spray

INTERVENTIONS:
Device: Fractional CO2 laser — Each patient will receive 6 sessions 2 weeks apart, after the laser treatment, a topical 5% minoxidil tincture will immediately applied.
  All patients will advised not to use any other treatment during the study
  Other Names: Drug
  Arms: Group 1
Device: Derma pen — , will be treated by microneedling using dermapen ( automated Derma Pen, DR Pen Ultima A6, China) which under complete aseptic precaution with a cartridge containing 12 needles moved diagonally, vertically, and horizontally for 4-5 times in each direction with 1.5 mm depth and speed 4-5(new cartridge every session), the application has been extended 1-2 cm perilesionally. The pinpoint bleeding will be considered an endpoint. topical 5% minoxidil tincture will immediately applied. Each patient will receive 6 sessions 2 weeks apart.
  Other Names: Drug
  Arms: Group 2
Drug: Niosome minoxidil — The patient of alopecia areata will be treated by topical nanominoxidil preparation twice daily for 3 months with no other treatment.
  Arms: Group 3
Drug: Minoxidil Topical Spray — The patient of alopecia areata will be treated by topical minoxidil 5% preparation twice daily for 3 months with no other treatment.
  Arms: Group 4

SUMMARY:
* Compare the clinical efficacy, and safety of transepidermal drug delivery of fractional CO2 laser versus microneedling followed by minoxidil 5% application for the treatment of alopecia areata.
* Evaluate the efficacy, and safety of minoxidil nanoparticles as a topical treatment of alopecia areata.

DETAILED DESCRIPTION:
Alopecia areata (AA) is the most common cause of non-scarring alopecia. (Hordinsky, 2013).

Although many patients improve spontaneously or respond to standard therapy, in patients with more severe and refractory disease, management can be quite challenging (Messenger et al., 2012 and Kranseler and Sidbury, 2017).

Corticosteroids either topical or intralesional are the most popular medications used to treat this condition. Other therapies such as topical minoxidil (MXD), anthralin, immunotherapy, systemic corticosteroids are also commonly used with variable success (Shumez et al., 2015).

Patients treated with MXD 5% have significant hair growth than placebo. Minoxidil was more effective for patchy alopecia than other types of AA such as ophiasis and alopecia totalis. It was ineffective in alopecia universalis (El-Taib et al., 2017).

In contrast, the incidence of adverse events associated with 10% MXD treatment was higher than with 5% MXD treatment. Therefore, new approaches are required to achieve both expected efficacy and safety (Oaku et al., 2022).

The combination of non-ablative laser and topical MXD can be a good alternative therapy for AA patients, including alopecia totalis and alopecia universalis, without systemic and local side effects (Wang et al., 2019) According to follicle deposition and diffusion experiments, minoxidil nanoemulsions penetrated hair follicles 26 times more efficiently than standard treatment (Cardoso and Barradas, 2020).

To the best our knowledge no previous research studied the effect of nanominoxidil solution in treatment of AA except in animal or compare transepidermal drug delivery versus topical nanominoxidil.

ELIGIBILITY:
Inclusion Criteria:

* The study will include patients with alopecia areata

Exclusion Criteria:

* Children below 18 years , pregnant and lactating women . patients with chronic hepatic, hematological disorders or immunocompromised patients.

patient recieved any treatment for alopecia areata in the last 3 months before the study.

patients with extensive types (alopecia totalis, universalis and surface area >50%).

Ages: 10 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
Regrowth scale | 6 months
  0 score (regrowth < 10%) no response
  score (regrowth 11-25%) poor response score (regrowth 26-50%) fair response score (regrowth 51-75%) satisfactory response score (regrowth ≥ 75%) excellent response
Mcdonald Hull and Norris Regrowth Scale (by trichoscope | 6 months
  Grade 1 - Regrowth of vellus hair. Grade 2 - Regrowth of sparse pigmented terminal hair. Grade 3 - Regrowth of terminal hair with patches of alopecia with patches of alopecia 50-75% in SALT score.
  Grade 4 - Regrowth of terminal hair on scalp with patches of alopecia > 75% in SALT score.

IPD SHARING:
Plan to Share IPD: Yes